CLINICAL TRIAL: NCT03692949
Title: A Safety, Tolerability, and Pharmacokinetics Study of LY3451838 in Healthy Subjects
Brief Title: A Study of LY3451838 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17123; J1H-MC-LAJA (Other: Eli Lilly & Company)
Record Dates: First submitted 2018-10-01; First posted 2018-10-02 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- 25 milligram (mg) LY3451838 Part A (Experimental): 25 mg LY3451838 single dose administered intravenously (IV)
  Interventions: Drug: LY3451838
- 75 mg LY3451838 Part A (Experimental): 75 mg LY3451838 single dose administered IV.
  Interventions: Drug: LY3451838
- 250 mg LY3451838 Part A (Experimental): 250 mg LY3451838 single dose administered IV.
  Interventions: Drug: LY3451838
- 500 mg LY3451838 Part A (Experimental): 500 mg LY3451838 single dose administered IV.
  Interventions: Drug: LY3451838
- 1000 mg LY3451838 Part A (Experimental): 1000 mg LY3451838 single dose administered IV.
  Interventions: Drug: LY3451838
- 1500 mg LY3451838 Part A (Experimental): 1500 mg LY3451838 single dose administered IV.
  Interventions: Drug: LY3451838
- 250 mg LY3451838 Part B (Experimental): 250 mg LY3451838 single dose administered subcutaneously (SC).
  Interventions: Drug: LY3451838
- Placebo (Placebo Comparator): Placebo matching single dose administered IV in Part A or administered SC in Part B.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3451838 — Administered IV Part A
  Arms: 25 milligram (mg) LY3451838 Part A
Drug: LY3451838 — Administered IV Part A
  Arms: 75 mg LY3451838 Part A
Drug: LY3451838 — Administered IV Part A
  Arms: 250 mg LY3451838 Part A
Drug: LY3451838 — Administered IV Part A
  Arms: 500 mg LY3451838 Part A
Drug: LY3451838 — Administered IV Part A
  Arms: 1000 mg LY3451838 Part A
Drug: LY3451838 — Administered IV Part A
  Arms: 1500 mg LY3451838 Part A
Drug: LY3451838 — Administered SC Part B
  Arms: 250 mg LY3451838 Part B
Drug: Placebo — Administered IV in Part A and SC in Part B
  Arms: Placebo

SUMMARY:
The study has two parts. In Part A, single increasing doses of LY3451838 will be administered intravenously (into a vein). In Part B, a single dose of LY3451838 will be administered subcutaneously (just under the skin).

ELIGIBILITY:
Inclusion Criteria:

* Male participants must adhere to contraception restrictions
* Female participants must be of non-childbearing potential due to:

  * Menopause: spontaneous amenorrhea for at least 12 months not induced by a medical condition such as anorexia nervosa and not taking medications that induced the amenorrhea (e.g., oral contraceptives, hormones, gonadotropin releasing hormone, anti-estrogens, selective estrogen receptor modulators, or chemotherapy)
  * Surgical sterilization
* Have a body mass index of 18 to 35 kilograms per square meter (kg/m²)
* Have clinical laboratory test results within normal reference range or with acceptable deviations
* Have an estimated glomerular filtration rate greater than or equal to (≥) 60 milliliters per minute per 1.73 meters squared (mL/minute/1.73 m²) of body surface area
* Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

* Are currently enrolled in or discontinued from a clinical trial within the last 30 days, or have previously completed or withdrawn from this study
* Have a history or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, renal, endocrine, psychiatric or neurological disease, or any clinically significant laboratory abnormality
* Have history of or presence of uncontrolled asthma, significant atopy, or significant rheumatological or autoimmune diseases
* Have had lymphoma, leukemia, or any malignancy within the past 5 years, or breast cancer within the past 10 years (with some exceptions)
* Have used, or intend to use some prescription or over the counter medications, including herbal medications within 14 days prior to dosing
* Have an abnormality in the 12-lead electrocardiogram (ECG) or Fridericia's corrected QT (QTcF)
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies, hepatitis C and/or positive hepatitis C antibody, or hepatitis B and/or positive hepatitis B surface antigen
* Have donated blood of more than 450 milliliters (mL) within the last 3 months
* Are unwilling to stop alcohol consumption while resident in the Clinical Research Unit (CRU)
* Have an average weekly alcohol intake that exceeds 21 units per week for males and 14 units per week for females (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Current smoker of more than 10 cigarettes or equivalent per day and unable to stop smoking while in the CRU
* Have an abnormal blood pressure
* Have clinically significant proteinuria or hematuria
* Positive findings for known drugs of abuse
* Have received treatment with biologic agents within 3 months or 5 half-lives (whichever is longer)
* Have clinically significant allergies, or intolerance to corticosteroids, or severe post treatment hypersensitivity reactions

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson MP, Krikke-Workel J, Patel CN, Morin SM, Turner PK, Clark KA, Donley D, Jin Y, Johnson KW, Vincent M, Stille JR, Broad LM, Patel A. Preclinical and clinical evaluation of LY3451838, a PACAP-neutralizing monoclonal antibody, in randomized, double-blind, placebo-controlled phase 1 and phase 2 studies involving healthy adults and adults with treatment-resistant migraine. Cephalalgia. 2025 Aug;45(8):3331024251368757. doi: 10.1177/03331024251368757. Epub 2025 Aug 21. PMID 40836866

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matching single dose administered IV in Part A and administered SC in Part B.
Period: Overall Study
Arm/Group | 25 Milligram (mg) LY3451838 Part A | 75 mg LY3451838 Part A | 250 mg LY3451838 Part A | 500 mg LY3451838 Part A | 1000 mg LY3451838 Part A | 1500 mg LY3451838 Part A | 250 mg LY3451838 Part B | Placebo
Started | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 14
Received at Least One Dose of Study Drug | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 14
Completed | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 Milligram (mg) LY3451838 Part A | 75 mg LY3451838 Part A | 250 mg LY3451838 Part A | 500 mg LY3451838 Part A | 1000 mg LY3451838 Part A | 1500 mg LY3451838 Part A | 250 mg LY3451838 Part B | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 14 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (10.1) | 44.0 (14.3) | 41.4 (14.1) | 40.2 (15.0) | 38.4 (9.6) | 43.3 (11.3) | 49.8 (6.0) | 40.5 (11.0) | 42.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 8
  Male | 3 | 4 | 5 | 6 | 5 | 6 | 4 | 12 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 5 | 5 | 6 | 5 | 6 | 6 | 14 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 14 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 14 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment Emergent Adverse Event
Description: A summary of other non-serious Adverse Events (AE's), and all Serious Adverse Events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through 20 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 Milligram (mg) LY3451838 Part A | 75 mg LY3451838 Part A | 250 mg LY3451838 Part A | 500 mg LY3451838 Part A | 1000 mg LY3451838 Part A | 1500 mg LY3451838 Part A | 250 mg LY3451838 Part B | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 14
Participants | 4 | 5 | 4 | 6 | 4 | 5 | 4 | 12

2. Primary Outcome: Number of Participants With One or More Serious Adverse Events
Description: A summary of other non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through 20 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 Milligram (mg) LY3451838 Part A | 75 mg LY3451838 Part A | 250 mg LY3451838 Part A | 500 mg LY3451838 Part A | 1000 mg LY3451838 Part A | 1500 mg LY3451838 Part A | 250 mg LY3451838 Part B | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Serum Concentration-Time Curve From 0 to Infinity (AUC 0 -∞) of LY3451838
Description: PK: AUC of LY3451838
Time Frame: Part A: Predose, End of Infusion, 3, 6, 12, 24, 36, 48 h, and Days 5, 7, 9, 15, 22, 29, 43, 57, 71, 85, and 141 post-dose; Part B: Predose, 3, 6, 12, 24, 36, 48 h, and Days 5, 7, 9, 15, 22, 29, 43, 57, 71, 85, and 141 post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg*h/mL)
Groups:
- 25 mg LY3451838 Part A: 25 mg LY3451838 single dose administered IV.
- 1000 mg LY3451838: 1000 mg LY3451838 single dose administered IV.
- 250 mg LY3451838 Part B: 250 mg LY3451838 single dose administered SC.
Arm/Group | 25 mg LY3451838 Part A | 75 mg LY3451838 Part A | 250 mg LY3451838 Part A | 500 mg LY3451838 Part A | 1000 mg LY3451838 | 1500 mg LY3451838 Part A | 250 mg LY3451838 Part B
Number analyzed (Participants) | 4 | 6 | 5 | 6 | 5 | 6 | 4
microgram*hour per milliliter (μg*h/mL) | 1580 (25.0) | 7510 (24.4) | 21900 (25.0) | 46100 (15.4) | 85500 (19.6) | 128000 (12.2) | 2040 (57.0)

4. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of LY3451838
Description: PK: Cmax of LY3451838
Time Frame: as for outcome 3
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | 25 mg LY3451838 Part A | 75 mg LY3451838 Part A | 250 mg LY3451838 Part A | 500 mg LY3451838 Part A | 1000 mg LY3451838 | 1500 mg LY3451838 Part A | 250 mg LY3451838 Part B
Number analyzed (Participants) | 4 | 6 | 5 | 6 | 5 | 6 | 6
microgram per milliliter (μg/mL) | 8.54 (39.1) | 30.9 (13.4) | 89.1 (15.8) | 172 (27.1) | 318 (24.1) | 523 (22.4) | 1.97 (113.7)

ADVERSE EVENTS:
Time Frame: Baseline up to 20 Weeks
Description: All participants who received at least one dose of study drug.
Groups:
- 25 mg LY3451838 Part A: 25 milligrams (mg) LY3451838 single dose administered Intravenously (IV).
- 250 mg LY3451838 Part B: 250 mg LY3451838 or Placebo administered subcutaneously (SC).
- Placebo: Placebo administered IV in Part A and administered SC in Part B.
Arm/Group | 25 mg LY3451838 Part A | 75 mg LY3451838 Part A | 250 mg LY3451838 Part A | 500 mg LY3451838 Part A | 1000 mg LY3451838 Part A | 1500 mg LY3451838 Part A | 250 mg LY3451838 Part B | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/6 | 0/5 | 0/6 | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/6 | 0/5 | 0/6 | 0/6 | 0/14
Other Adverse Events (participants affected / at risk) | 4/5 | 5/6 | 4/5 | 6/6 | 4/5 | 5/6 | 4/6 | 12/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg LY3451838 Part A (N=5) | 75 mg LY3451838 Part A (N=6) | 250 mg LY3451838 Part A (N=5) | 500 mg LY3451838 Part A (N=6) | 1000 mg LY3451838 Part A (N=5) | 1500 mg LY3451838 Part A (N=6) | 250 mg LY3451838 Part B (N=6) | Placebo (N=14)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Catheter site paraesthesia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Vessel puncture site bruise (General disorders) | 2 (3) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 4 (5)
Vessel puncture site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 2 (5) | 2 (3) | 2 (4)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03692949/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03692949/SAP_001.pdf